CLINICAL TRIAL: NCT06722664
Title: A Phase 2 , Randomized, Placebo-Controlled, Double-Blind Study to Evaluate the Safety and Efficacy of Using Premedication With OsrhCT and Dimethicone Emulsion During Upper Gastrointestinal Endoscopy Examination.
Brief Title: Efficacy and Safety of OsrhCT and Dimethicone Emulsion Before Upper Endoscopy on Visualization of the Gastric Mucosa.
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Healthgen Biotechnology Corp. (Industry)
Collaborators: Beijing Friendship Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Diagnostic
Other Study IDs: HY1005-1-2024-P2
Record Dates: First submitted 2024-11-26; First posted 2024-12-09 (Actual); Last update posted 2025-04-29 (Actual); Status verified 2024-12

CONDITIONS: Gastric Mucosal Lesion
Keywords: OsrhCT; Recombinant Human Chymotrypsin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Recombinant Human Chymotrypsin(OsrhCT) 4000U (Experimental)
  Interventions: Drug: Recombinant Human Chymotrypsin(OsrhCT) 4000U; Drug: Placebo for Recombinant Human Chymotrypsin(OsrhCT); Drug: Dimethicone emulsion 4ml
- Recombinant Human Chymotrypsin(OsrhCT) 8000U (Experimental)
  Interventions: Drug: Recombinant Human Chymotrypsin(OsrhCT) 4000U; Drug: Dimethicone emulsion 4ml
- Placebo for Recombinant Human Chymotrypsin(OsrhCT) (Placebo Comparator)
  Interventions: Drug: Placebo for Recombinant Human Chymotrypsin(OsrhCT); Drug: Dimethicone emulsion 4ml

INTERVENTIONS:
Drug: Recombinant Human Chymotrypsin(OsrhCT) 4000U — Recombinant Human Chymotrypsin (OsrhCT), provided by Wuhan Healthgen Biotechnology Corporation, 4,000U/vial, freeze-dried powder
  Arms: Recombinant Human Chymotrypsin(OsrhCT) 4000U; Recombinant Human Chymotrypsin(OsrhCT) 8000U
Drug: Placebo for Recombinant Human Chymotrypsin(OsrhCT) — Recombinant Human Chymotrypsin (OsrhCT), provided by Wuhan Healthgen Biotechnology Corporation, 0 U/vial, freeze-dried powder
  Arms: Placebo for Recombinant Human Chymotrypsin(OsrhCT); Recombinant Human Chymotrypsin(OsrhCT) 4000U
Drug: Dimethicone emulsion 4ml — Dimethicone emulsion，produced by Sichuan Jian Neng Pharmaceutical Co., Ltd, 6ml/bottle.

SUMMARY:
Study was designed to evaluate efficacy of OsrhCT and Dimethicone emulsion before upper endoscopy on visibility of gastric mucosa.

A total of 336 subjects (both male and female) are expected to be enrolled in this trial.

DETAILED DESCRIPTION:
This is a monocentric, double-blind, randomized study involving 336 patients indicated for diagnostic upper endoscopy. Patients were randomly assigned to one of three arms, with OsrhCT 4000U+ Dimethicone emulsion 4ml , with OsrhCT 8000U+ Dimethicone emulsion 4ml , and with placebo for OsrhCT+ Dimethicone emulsion 4ml. During the examination, each photograph was individually taken in 5 defined areas. The first 30 cases were collected to establish standards and method validation. The visibility score was given by the sum of the score 1-4 from 5 defined localities evaluated by a blinded endoscopist and subsequently by two or three blinded endoscopists. Other parameters monitored were examination time and a semiquantitative evaluation of residual gastric fluid.

ELIGIBILITY:
Inclusion Criteria:

1. Patients indicated for gastroscopy examination;
2. Subjects fully understand the content, process, and possible adverse reactions of the trial and voluntary participation with signed informed consent;
3. Able to complete the research according to the requirements of the experimental plan;
4. Subjects (including their spouses) voluntarily have no pregnancy plans and use contraception during the study and within 3 months after the last administration of the study drug;
5. Aged 18-75 years (inclusive), male or female;

Exclusion Criteria:

1. Known allergy to chymotrypsin; Known to be allergic to preparation or anesthesia medication before gastroscopy examination;
2. Patients plan to undergo gastroscopic treatment, such as endoscopic titanium clip for hemostasis, esophagogastric fundal variceal ligation, endoscopic mucosal stripping, etc;
3. Subjects accessed not to stand sedation anesthesia or gastroscopy examination;
4. Severe cardiovascular, pulmonary, or cerebral diseases, such as angina, heart failure, and new-onset stroke; or severe liver disease, cirrhosis, or esophagogastric fundus varices;
5. Suspected or known esophageal fistula, tracheal fistula, intestinal obstruction, active gastrointestinal bleeding, gastric perforation, history of anatomically altered upper GI surgery;
6. Abnormal laboratory values:: alanine aminotransferase (ALT)>2 × ULN, aspartate aminotransferase (AST)>2 × ULN, serum creatinine>1.5 × ULN;
7. Female subjects who had unprotected sex within 14 days prior to screening;
8. Pregnant or breastfeeding women;
9. Subjects who have participated in any drug clinical trial and received treatment within the last 3 months;
10. Any other conditions deemed unsuitable for the study by the investigator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 336 (Estimated)
Dates: Start 2024-12-19 (Actual); Primary Completion 2025-05-15 (Estimated); Study Completion 2025-05-15 (Estimated)

PRIMARY OUTCOMES:
Total visibility score (TVS) evaluated by blinded endoscopists | Through study completion, an average of 3 months
  "Total visibility score"counted as the sum of visibility score in lower esophagus, gastric fundus, upper gastric body, lower gastric body and gastric antrum.

SECONDARY OUTCOMES:
Vsibility scores evaluated by blinded endoscopists for mucosain of 5 various anatomical parts of the stomach | Through study completion, an average of 3 months
  Vsibility scores for the lower esophagus, antrum, lower gastric body, upper gastric body, and fundus.
The amount of water flushed for satisfactory observation of the upper gastrointestinal tract | during diagnostic upper endoscopy, up to 1 hour
  Amount of water used to allow an suitable visualization of gastric mucosa
Duration of endoscopy | during diagnostic upper endoscopy, up to 1 hour
  Time to complete the upper endoscopy (from the time of oral intubation until complete removal of the endoscope)
Incidence of adverse events | up to 1 week
  Number of gastroscopy procedures with adverse event divided by the number of all gastroscopy procedures. Number of participants with treatment-related adverse events as assessed by CTCAE V5.0.

OTHER OUTCOMES:
Establishment and method validation of the criteria for mucosal visibility score | Through study completion, an average of 3 months
  The first 30 cases were collected to establish standards and method validation. The visibility score was given by the sum of the score 1-4 from 5 defined localities (lower esophagus, gastric fundus, upper gastric body, lower gastric body and gastric antrum) evaluated by a blinded endoscopist and subsequently by two or three blinded endoscopists.

CONTACTS AND LOCATIONS:
Overall Officials: Shutian Zhang, MD, Principal Investigator — Beijing Friendship Hospital; Fandong Meng, MD, Principal Investigator — Beijing Friendship Hospital
Locations (5):
- China (5):
  - Beijing Friendship Hospital, Beijing, Beijing Municipality
  - Chinese PLA Central Theatre General Hospital, Wuhan, Hubei
  - Renmin Hospital of Wuhan University, Wuhan, Hubei
  - the Central Hospital of Wuhan, Wuhan, Hubei
  - Inner Mongolia Autonomous Region People's Hospital, Hohhot, Inner Mongolia

IPD SHARING:
Plan to Share IPD: No